CLINICAL TRIAL: NCT00717652
Title: Efficiency And Safety Of Association Arbutin, Triamcinolone And Tretinoin In The Treatment Of Facial Melasma, Taking As Reference The Product Triluma ® (Hidroquinone, Fluoncinolone And Tretinoin).
Brief Title: Efficiency And Safety Of Association Arbutin, Triamcinolone And Tretinoin In Treatment Of Melasma
Acronym: melasma
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATTGLE0508
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Arbutin; Tretinoin; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): arbutin, tretinoin, triamcinolone
  Interventions: Drug: arbutin, tretinoin, triamcinolone
- 2 (Active Comparator): Triluma
  Interventions: Drug: Triluma

INTERVENTIONS:
Drug: arbutin, tretinoin, triamcinolone — arbutin, tretinoin, triamcinolone
  Arms: 1
Drug: Triluma — Hydroquinone, Fluoncinolone, Tretinoin
  Arms: 2

SUMMARY:
The objective of this study is evaluating the clinical activity of the association (tretinoin + arbutin + triamcinolone) in the treatment of epidermal melasma.

DETAILED DESCRIPTION:
The melasma is a common hipermelanosis, acquired, symmetrical, with irregular occurring in areas such as photo-exposed face, forehead and temples, can affect the eyelids and tion. The facial regions most affected are: zigomatic (82.4%), parotid (64.7%), front (64.7%), mandible (35.3%) and nasal (35.3%). The injuries of melasma is variable increase of epidermal melanin and inflammatory infiltrate of mild to moderate intensity. Treatment with compounds such as hydroquinone and derivatives, tretinoin, corticosteroids moderate or combination of them all have shown good results, diminishing the training, reducing the stability and promoting the destruction of melanocytes. The primary objective of this study is evaluating the clinical activity of the association (tretinoin + arbutin + triamcinolone) manufactured by Glenmark Laboratory, and as the comparator drug product Triluma ® (hydroquinone + fluocinolone + tretinoin), in the treatment of epidermal melasma through parameters of clinical course of the disease (improves) and its security.

Patients who are included in the study will be randomly and automatically receive one of the treatments (New association or Triluma ®), which should use for 12 weeks. The products should be applied in the regions affected once a day, during night.

The evaluation of clinical improvement, as well as security, will be held on periodic visits, as described below, which will be held the record and supply of medicines to patients.

In each visit, beyond the clinical examination of photographs and large, it filled the Area and Severity Scale (Melasma Area and Severity Index - MASI), which quantifies the melasma and will be the main tool of control of clinical improvement.

At the end of the study, data will be compared, showing no inferiority or inferiority of clinical drug testing in relation to the comparator.

ELIGIBILITY:
Inclusion Criteria:

* Women adults aged more than 18 years;
* Patients suffering from melasma Epidermal the face of mild and moderate;
* Patients who have not done any treatment for melasma in the 3 months preceding the study;
* Patients with good mental and physical health;
* Patients who agree with the purposes of the study and sign the TCLE.

Exclusion Criteria:

* Patients with skin diseases other than melasma, which interfere in clinical evaluation as hemangiomas and queloides;
* Patients with melasma skin or mixed;
* Patients with sensitivity to agents hipopigmentantes;
* Patients with sensitivity to fotoprotetores;
* Patients who are pregnant or breastfeeding;
* Patients who, at the discretion doctor, are not able to participate in the study;
* Patients who have carried out any treatment for melasma in the 3 months preceding the study
* Patients who do not agree with the terms described in the Statement of Informed Consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-07 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07

PRIMARY OUTCOMES:
evaluating the clinical activity of the association (tretinoin + arbutin + triamcinolone)in the treatment of epidermal melasma. | arbutin triamcinolone tretinoin

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, S, Brazil